CLINICAL TRIAL: NCT05410886
Title: A Questionnaire-based Study to Improve the Diagnosis of Functional Hypothalamic Amenorrhea (FHA) in Women With Secondary Amenorrhea Attending Hospital
Brief Title: Screening Women for Functional Hypothalamic Amenorrhea (FHA)
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 20HH6115
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Amenorrhea Secondary
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — A questionnaire including up to 20 questions will be distributed to study participants. This questionnaire will be used to identify women with FHA.

SUMMARY:
What do the investigators know already? Many women suffer loss of periods (amenorrhoea). One of the most common causes of period loss is called 'functional hypothalamic amenorrhea' (FHA). FHA is difficult to diagnose and may be mistaken for other conditions causing period loss, such as polycystic ovarian syndrome (PCOS). This could cause delays in starting the correct treatment.

What is the justification for doing this study? Undiagnosed women with FHA are predisposed to complications related to low oestrogen levels, such as osteoporosis, bone fractures and infertility. The failure to accurately identify women with FHA and mislabel those women with FHA as having PCOS, may delay appropriate treatment. Treatment delay causes harm for affected women, including bone fractures and infertility.

What do the investigators propose? Improve the diagnosis of women with FHA by composing an assessment score, which could be used by women to improve the accuracy of diagnosing FHA. The investigators designed a questionnaire based on literature search, which can be used to identify women with FHA. A questionnaire-based study (on-line or in person) will be performed to identify risk of FHA, in women referred to hospital with period loss.

DETAILED DESCRIPTION:
A questionnaire was developed to be used by women with period loss to facilitate the diagnosis of women with FHA. The development of the questionnaire was based on systematic literature review and comments from a small patient involvement group, as per National Institute for Health and Care Research (NIHR) INVOLVE guidelines.

Participants will be recruited via distributing a patient information sheet, consent form and a questionnaire to all women referred with amenorrhea to the Endocrinology or Reproductive Medicine clinics at Imperial College Healthcare NHS Trust and/or participating NHS organisations. Completion of the consent form and questionnaire is entirely dependent on each potential participant's choice.

Every woman taking part can complete the questionnaire before or after her appointment. All questionnaires will be anonymised with a unique study code, and handed back to the NHS clinician.

ELIGIBILITY:
Inclusion Criteria:

* Any woman 18-58 years of age
* Secondary amenorrhea defined by either menstrual cycle interval persistently exceeding 45 days and/or those with period loss for 3 months or more

Exclusion Criteria:

* Women who never had periods (primary amenorrhea).

Ages: 18 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women referred by their GP with amenorrhea to the Endocrinology or Reproductive Medicine clinics at Imperial College Healthcare NHS Trust hospitals and participating NHS organisations.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Frequency of clinical features in women with Functional hypothalamic amenorrhea | 3 years
  Descriptive statistics will be applied to questionnaire responses looking at frequency of different clinical features in women with FHA and women with other diagnoses.

OTHER OUTCOMES:
Frequency of biochemical features in women with Functional hypothalamic amenorrhea | 3 years
  Descriptive statistics will be applied to standard medical investigation results looking at frequency of different biochemical features in women with FHA and women with other diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Channa Jayasean, PhD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - University College London Hospital NHS Trust, London
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Background] Phylactou M, Clarke SA, Patel B, Baggaley C, Jayasena CN, Kelsey TW, Comninos AN, Dhillo WS, Abbara A. Clinical and biochemical discriminants between functional hypothalamic amenorrhoea (FHA) and polycystic ovary syndrome (PCOS). Clin Endocrinol (Oxf). 2021 Aug;95(2):239-252. doi: 10.1111/cen.14402. Epub 2021 Jan 19. PMID 33354766
- [Result] Abou Sherif S, Newman R, Haboosh S, Al-Sharefi A, Papanikolaou N, Dimakopoulou A, Webber LJ, Abbara A, Franks S, Dhillo WS, Jayasena CN. Investigating the potential of clinical and biochemical markers to differentiate between functional hypothalamic amenorrhoea and polycystic ovarian syndrome: A retrospective observational study. Clin Endocrinol (Oxf). 2021 Oct;95(4):618-627. doi: 10.1111/cen.14571. Epub 2021 Aug 9. PMID 34323305